CLINICAL TRIAL: NCT04712435
Title: Prospective, Randomized Study Using N-Acetylcysteine as Prophylaxis of Sinusoidal Obstruction Syndrome in Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy of N-acetylcysteine Versus Placebo as Prophylaxis of Sinusoidal Obstruction Syndrome in Patients Undergoing Hematopoietic Stem Cell Transplantation
Acronym: ALISON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Principal Investigator, Jamilla Neves Cavalcante, Principal Investigator, Instituto Brasileiro de Controle do Cancer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 33788420.4.0000.0072
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-01

CONDITIONS: Sinusoidal Obstruction Syndrome (SOS); Hematopoietic Stem Cell Transplant (HSCT)
Keywords: Stem cell transplant; Hematopoietic stem cell transplant (HSCT); Sinusoidal obstruction syndrome (SOS); Veno-occlusive disease (VOD); N-acetylcysteine
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This is a single-center, randomized, placebo-controlled study to evaluate the efficacy and safety of N-acetylcysteine
Who Masked: Participant, Investigator
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: N-acetylcysteine (Experimental): Sachets containing N-acetylcysteine 200 mg Powder for Oral Solution administered every 8 hours (Daily dose 600 mg/day). is administered on the first day of conditioning and will continue until Day +30 post HSCT or hospital discharge, whichever is sooner
  Interventions: Drug: N-acetylcysteine
- Placebo Comparator: Placebo (Placebo Comparator): 200mg granulated solution of matching placebo administered every 8 hours (Daily dose 600 mg/day), is administered on the first day of conditioning and will continue until Day +30 post HSCT or hospital discharge, whichever is sooner
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Eligible patients will be randomised to receive N-acetylcysteine versus matching placebo
  Arms: Experimental: N-acetylcysteine
Drug: Placebo — Eligible patients will be randomised to receive N-acetylcysteine versus matching placebo
  Arms: Placebo Comparator: Placebo

SUMMARY:
Sinusoidal obstruction syndrome (SOS) or hepatic veno-occlusive disease (VOD) is a serious complication that occurs, most often occurring in patients undergoing hematopoietic stem cell transplantation (HSCT), especially in its first thirty days. The morbidity and mortality in this syndrome are considerable, since severe SOS is associated with a mortality of more than 90% in the first hundred days of HSCT.

Some risk factors are modifiable, especially those related to transplantation, but when non-alterable factors are present, preventive measures are needed that can reduce the incidence and / or severity of SOS.

DETAILED DESCRIPTION:
This is a single-center, randomized, placebo-controlled study to evaluate the efficacy and safety of N-acetylcysteine as prophylaxis of sinusoidal obstruction syndrome in patients undergoing hematopoietic stem cell transplantation Up to date, no approved medications are available for prophylactic treatment of sinusoidal obstruction syndrome in patients undergoing hematopoietic stem cell transplantation. N-acetylcysteine is a drug that has been long used as a mucolytic. And placebo responses contribute to help assess the appropriateness of randomized clinical trials in determining the size of drug effect.

The study will enroll patients undergoing hematopoietic stem cell transplantation to receive sequentially one of two treatment: N-acetylcysteine or Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age ≥ 18 years
* A proven diagnosis of one of the hematological malignancies: Acute Myeloid Leukemia, Acute Lymphoid Leukemia, Chronic Myeloid Leukemia, Chronic Lymphoid Leukemia, Multiple Myeloma, Non-Hodgkin's Lymphoma, Hodgkin's Lymphoma
* Patients must be scheduled to undergo of Allogeneic hematopoietic transplantation or HLA (Human Leukocyte Antigen) haploidentical related or Unrelated or HLA-matched related or autologous stem cell transplant
* Patients must be able to understand and sign a written informed consent

Exclusion Criteria:

* Patient has a serious active disease or co-morbid medical condition, as judged by the investigator, which would interfere with the conduct of this study
* Patient, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
* Known hypersensitivity to N-acetylcysteine
* Contraindications to perform any procedure provided for in this study
* Patients who have already undergone a previous transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of SOS | Day + 30 post HSCT
  To evaluate if prophylactic of N-acetylcysteine has an impact on the incidence of Sinusoidal obstruction syndrome (SOS)

SECONDARY OUTCOMES:
Severity of SOS | within 30 days of bone marrow transplant
  Death as noted in medical record
Sinusoidal obstruction syndrome (SOS) -Free Survival at Day 30 Post-Hematopoietic Stem Cell Transplant (HSCT) | 30 Days Post-Transplant
  Comparison of efficacy of N-acetylcysteine vs Placebo for the prevention of SOS

CONTACTS AND LOCATIONS:
Overall Officials: Jamilla N Cavalcante, MD, Principal Investigator — IBCC Oncologia
Locations (1):
- Jamilla Neves Cavalcante, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dignan FL, Wynn RF, Hadzic N, Karani J, Quaglia A, Pagliuca A, Veys P, Potter MN; Haemato-oncology Task Force of British Committee for Standards in Haematology; British Society for Blood and Marrow Transplantation. BCSH/BSBMT guideline: diagnosis and management of veno-occlusive disease (sinusoidal obstruction syndrome) following haematopoietic stem cell transplantation. Br J Haematol. 2013 Nov;163(4):444-57. doi: 10.1111/bjh.12558. Epub 2013 Sep 17. PMID 24102514
- [Background] Mohty M, Malard F, Abecassis M, Aerts E, Alaskar AS, Aljurf M, Arat M, Bader P, Baron F, Bazarbachi A, Blaise D, Ciceri F, Corbacioglu S, Dalle JH, Duarte RF, Fukuda T, Huynh A, Masszi T, Michallet M, Nagler A, NiChonghaile M, Pagluica T, Peters C, Petersen FB, Richardson PG, Ruutu T, Savani BN, Wallhult E, Yakoub-Agha I, Carreras E. Sinusoidal obstruction syndrome/veno-occlusive disease: current situation and perspectives-a position statement from the European Society for Blood and Marrow Transplantation (EBMT). Bone Marrow Transplant. 2015 Jun;50(6):781-9. doi: 10.1038/bmt.2015.52. Epub 2015 Mar 23. PMID 25798682
- [Background] Dalle JH, Giralt SA. Hepatic Veno-Occlusive Disease after Hematopoietic Stem Cell Transplantation: Risk Factors and Stratification, Prophylaxis, and Treatment. Biol Blood Marrow Transplant. 2016 Mar;22(3):400-9. doi: 10.1016/j.bbmt.2015.09.024. Epub 2015 Oct 23. PMID 26431626
- [Background] Ozdemir ZC, Turhan AB, Eren M, Bor O. Is N-acetylcysteine infusion an effective treatment option in L-asparaginase associated hepatotoxicity? Blood Res. 2017 Mar;52(1):69-71. doi: 10.5045/br.2017.52.1.69. Epub 2017 Mar 27. No abstract available. PMID 28401107
- [Background] Barkholt L, Remberger M, Hassan Z, Fransson K, Omazic B, Svahn BM, Karlsson H, Brune M, Hassan M, Mattsson J, Ringden O. A prospective randomized study using N-acetyl-L-cysteine for early liver toxicity after allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 May;41(9):785-90. doi: 10.1038/sj.bmt.1705969. Epub 2008 Jan 7. PMID 18176610
- [Background] Ringden O, Remberger M, Lehmann S, Hentschke P, Mattsson J, Klaesson S, Aschan J. N-acetylcysteine for hepatic veno-occlusive disease after allogeneic stem cell transplantation. Bone Marrow Transplant. 2000 May;25(9):993-6. doi: 10.1038/sj.bmt.1702387. PMID 10800069